CLINICAL TRIAL: NCT05900531
Title: A 28-Day Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of K-757 in Healthy Overweight/Obese Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of K-757 in Healthy Overweight/Obese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-757 P004
Record Dates: First submitted 2023-04-07; First posted 2023-06-12 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- K-757 (Panel A) (Experimental)
  Interventions: Drug: K-757
- K-757 (Panel B) (Experimental)
  Interventions: Drug: K-757
- K-757 + sitaglipitin (Panel C) (Experimental)
  Interventions: Drug: K-757 and open-label sitagliptin
- K-757 and K-833 (Panel D) (Experimental)
  Interventions: Drug: K-757 and K-833
- K-757 and K-833 (Panel E) (Experimental)
  Interventions: Drug: K-757 and K-833
- Panel A (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757
- Panel B (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757
- Panel C (+ sitagliptin) (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757, open-label sitagliptin
- Panel D (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757 and matching placebo to K-833
- Panel E (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757 and matching placebo to K-833

INTERVENTIONS:
Drug: K-757 — administered orally
  Arms: K-757 (Panel A); K-757 (Panel B)
Drug: K-757 and open-label sitagliptin — both administered orally
  Arms: K-757 + sitaglipitin (Panel C)
Drug: Matching placebo to K-757 — administered orally
  Arms: Panel A; Panel B
Drug: Matching placebo to K-757 and matching placebo to K-833 — both administered orally
  Arms: Panel D; Panel E
Drug: K-757 and K-833 — both administered orally
  Arms: K-757 and K-833 (Panel D); K-757 and K-833 (Panel E)
Drug: Matching placebo to K-757, open-label sitagliptin — both administered orally
  Arms: Panel C (+ sitagliptin)

SUMMARY:
This is a multiple dose study to evaluate the safety, tolerability, PK, and PD of K-757 alone, in combination with sitagliptin, or in combination with K-833.

ELIGIBILITY:
Inclusion Criteria:

l. Understand the trial procedures and agree to participate by providing written informed consent.

2. Be willing and able to comply with all trial procedures and restrictions, including following study diet requirements.

3. Be healthy between 18 to 60 years of age, inclusive, at the Screening Visit.

4. Have a Body Mass Index (BMI) ≥27.0 and <35.0 (kg/m2) at the Screening Visit.

5. Be weight stable (<5% variation) over the last 3 months.

6. Be a nonsmoker who has not used tobacco or nicotine-containing products (e.g. nicotine patch, e-cigarettes, vapes) for at least 3 months before administration of the initial dose of trial drug and agrees to abstain from smoking tobacco or the use of nicotine-containing products while on study.

7. Be judged to be in good health by the Investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead ECG, and vital sign measurements performed at the Screening Visit and before administration of the initial dose of trial drug.

8. Meet the following requirements:

1. Is a male who agrees to all of the following:

   * To use an appropriate method of contraception, including a condom with or without spermicidal cream or jelly, from the first dose of study drug until 14 days after the last dose of study drug. A male subject who had a vasectomy procedure must follow the same restrictions as a non-vasectomized man.
   * If partner is pregnant, to use a condom
   * To not donate sperm from the first dose of study drug until 14 days after the last dose of study drug.

   OR
2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:

   * Postmenopausal (aged >45 years and with a minimum of 12 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level >30 mIU/mL).
   * Post hysterectomy, bilateral oophorectomy or bilateral salpingectomy, based on the subject's recall of their medical history.

Exclusion Criteria:

1. Has participated in another interventional investigational study within 30 days of the Screening Visit. The window will be derived from the date of the last study procedure and/or AE related to the study procedure in the previous study to the Screening Visit of the current study. If the subject received an investigational medication in the prior study, at least 5 half-lives (or longer if required by local regulations) must have passed between the last dose of the investigational product and the Screening Visit.
2. Is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the Sponsor or study site.
3. Has a history of multiple significant and/or any severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
4. Has a known hypersensitivity or contraindication to any component of K-757 (all Panels), sitagliptin (Panel C only), or K-833 (Panels D and E only), related compounds or their excipients.
5. Has a positive alcohol or drug screen at Screening or admission.
6. Has a positive pregnancy test.
7. Is a lactating/nursing female.
8. Has a positive test result for hepatitis B surface antigen (Ag), hepatitis C virus antibody, or human immunodeficiency (HIV) antibody, at the Screening Visit. Note: Subjects with positive hepatitis B virus or hepatitis C virus serology may be enrolled if quantitative polymerase chain reaction for hepatitis B virus or hepatitis C virus ribonucleic acid is negative.
9. Does not meet study site COVID-19 admission/study participation restrictions.
10. Has a fever (>38°C)*.
11. Had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit*.
12. Is unable to refrain from the use of prohibited prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication through completion of study participation. Allowable concomitant medications are limited to 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins), ≤2 permissible anti-hypertensive agents, and post-menopausal hormone replacement therapy (HRT). Statin doses must have been stable with reported compliance of at least 80% for ≥3 months prior to the Screening Visit. Anti-hypertensive and HRT doses/regimens must have been stable for ≥1 month prior to the Screening Visit.
13. Has been on any GLP-1 receptor agonist, any dipeptidyl peptidase IV (DPP-4) inhibitor, or any approved or investigational medications known to cause weight loss in the prior 3 months.
14. Has excessive consumption of alcohol within 6 months prior to screening (>14 drinks/week for men and >7 drinks/week for women, where l drink= 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) or use of soft drugs (such as marijuana) within 3 months prior to Screening, or hard drugs (such as cocaine) within 6 months prior to Screening.
15. Is unwilling or unable to refrain from consuming alcohol from 7 days prior to the first dose of study medication through the completion of study participation.
16. Is unable or unwilling to refrain from consumption of Seville oranges, grapefruit, grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids from 2 weeks prior to administration of the first dose of study drug, throughout the study, and until the Follow-up Visit.
17. Is unwilling to refrain from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard) or charbroiled meats beginning approximately 48 hours prior to admission to the clinic, if possible (if subject has consumed any of these items prior to admission, the subject may be included in the study and the food and amount should be recorded in the source documents). Subjects will not consume any of the above foods while in the clinical research unit and until the poststudy visit.
18. Has a substance abuse disorder.
19. Had a previous major psychotic disorder.
20. Has a corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec) for males and >470 msec for females at screening or on Day 1 predose.
21. Has a mean value for triplicate semi-recumbent systolic blood pressure >150 mmHg and/or diastolic blood pressure (BP) >90 mmHg measured after at least 10 minutes at rest at the Screening Visit.
22. Has a screening estimated glomerular filtration rate (eGFR by Modification of Diet in Renal Disease [MDRD]) <60 mL/min/1.73 m2.
23. Has alanine aminotransferase or aspartate aminotransferase (ALT or AST) of >1.0X upper limit of normal (ULN) or total bilirubin >1.2X ULN (isolated bilirubin >1.2X ULN is acceptable if bilirubin is fractionated and direct bilirubin is within the laboratory normal range) at the Screening Visit and Day -1. (Note: Subjects who do not meet this criterion during screening or check-in [Day -1] may not be rescreened/retested).
24. Has serum amylase or lipase >1.2X the ULN at the Screening Visit.
25. Has a recent history (within past 3 years) or current diagnosis of any of the following GI (gastro-intestinal) related diseases: intestinal obstruction, GI perforation, GI motility disorders, adhesions, Clostridium difficile colitis or have had recent unexplained GI bleeding within 3 months prior to screening.
26. Has any history of pancreatitis (acute or chronic), gastroparesis, ischemic colitis, inflammatory bowel disease (IBD), celiac disease, irritable bowel syndrome (IBS), or colitis.
27. Has any past surgical history of gastric banding or bariatric surgery or bowel resection.
28. Has a history of clinically significant endocrine disease including T2DM, a screening HbA1c ≥6.5%, or a history of clinically significant gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, neurologic disorder, neoplastic, or genitourinary abnormalities or diseases.
29. Has a history of unexplained arthralgias (Panel C only).
30. Has a history of bullous pemphigoid (Panel C only).
31. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

note-* Subject may be included if they are able to return to the site within 7 days of initial screening and the exclusion criterion is no longer met.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who experienced 1 or more treatment-emergent AEs | Up to Day 42 +/- 2 days
  after treatment with K-757 administered alone, when co-administered with sitagliptin, and when co-administered with K-833
Proportion of participants who discontinued study medication due to an AE | Up to Day 42 +/- 2 days
  after treatment with K-757 administered alone, when co-administered with sitagliptin, and when co-administered with K-833

SECONDARY OUTCOMES:
Area under the concentration-time curve [AUC] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
Maximum concentration [Cmax] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
Time of maximum concentration [Tmax] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
Clearance [Cl] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
Volume of distribution at steady-state [Vdss] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
Half-life [t1/2] of plasma K-757 | Days 1 and 28
  following multiple doses of K-757
AUC of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
Cmax of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
Tmax of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
Cl of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
Vdss of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
t1/2 of plasma K-757 | Days 1 and 28
  following multiple doses of K-757 when co-administered with sitagliptin
AUC of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Cmax of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Tmax of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Cl of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Vdss of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
t1/2 of plasma K-757 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
AUC of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Cmax of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Tmax of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Cl of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
Vdss of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833
t1/2 of plasma K-833 | Days 14 and 28
  following multiple doses of K-757 when co-administered with K-833

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States